CLINICAL TRIAL: NCT01876407
Title: Effectiveness of Low Energy Laser Treatment in Oral Mucositis Induced by Chemotherapy and Radiotherapy in Head and Neck Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FPS-LAS-2012-04; 001001006001 (Other Grant/Funding Number: AETSA)
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low energy laser (Experimental): Administration of a low energy laser for oral mucositis.
  Interventions: Device: Low intensity laser for oral mucositis
- Placebo (Placebo Comparator)
  Interventions: Device: Low intensity laser for oral mucositis switch off

INTERVENTIONS:
Device: Low intensity laser for oral mucositis
  Arms: Low energy laser
Device: Low intensity laser for oral mucositis switch off — Low intensity laser for oral mucositis switch off
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of using to low intensity laser as an intervention against preventive and therapeutic oral mucositis induced by radiotherapy and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with squamous cell carcinoma of the oral cavity.
* Patients aged between 18 and 80 years.
* Patients who are to receive one of the following treatment
* Combined radiotherapy (conventional fractionation 70 Gy reaching the tumor and affected lymph nodes, and 50 Gy in the areas ganglion drainage) and chemotherapy (cisplatin 100 mg/m2 IV on days 1, 22 and 43 irradiation or cetuximab 400mg/m2 as a single dose pre-load radiotherapy and 250mg/m2 weekly for the same. Regardless of whether they have received previous surgical treatment.
* Treatment with radiotherapy of 70 Gy in 35 daily sessions 2Gy/día consecutive.
* Patients who voluntarily express their intention to participate by informed consent.

Exclusion Criteria:

* Patients who denied informed consent.
* Patients who have hypersensitivity or allergy to any of the components included in the study.
* Patients diagnosed with HIV, and autoimmune diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of using low-intensity laser compared with placebo as preventive and therapeutic intervention of oral mucositis induced by radiation therapy and chemotherapy. | 24 months

SECONDARY OUTCOMES:
Evaluate the effectiveness of using low level laser compared with placebo in the prevention of onset of oral mucositis induced by treatment of head and neck QRT. | 24 months
Evaluate the effectiveness of the use of low laser intensity versus placebo in improving the healing of oral mucositis induced by treatment of head and neck QRT. | 24 months
Evaluate the effectiveness of using low level laser compared with placebo in reducing pain during and after cancer treatment. | 24 months
Evaluate the effectiveness of using low level laser compared with placebo in analgesic use during and after cancer treatment. | 24 months
Assess the intervention tolerance and side effects of it. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Torres Lagares, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Spain